CLINICAL TRIAL: NCT06775301
Title: Dispersed Clinical Validation of the Hyfe Cough Monitoring System
Status: Completed | Type: Observational
Sponsor: Hyfe Inc (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: ID206-2
Record Dates: First submitted 2025-01-13; First posted 2025-01-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cough Frequency
Keywords: Cough monitoring
MeSH Terms: conditions — Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Hyfe Cough Monitoring System — Smartwatch-based cough monitoring

SUMMARY:
This study will test the accuracy of the Hyfe Cough Monitoring System. This system uses a smartwatch to record the number and pattern of coughs (like a "Fitbit for cough").

The investigators will compare the coughs counted by the Hyfe device with manual cough counts from environmental sounds recordings in the same period.

This is a dispersed observational study and will include individuals with a variety of cough related conditions including but not limited to refractory or unexplained cough, Bronchiectasis, COPD, COVID-19, non-tuberculous mycobacterial infection, tuberculosis, or upper respiratory tract infection.

DETAILED DESCRIPTION:
The Hyfe Cough Monitoring System is investigational, which means that it has not been approved by the Food and Drug Administration (FDA). This study is funded by Hyfe, Inc. and executed under the direction of Dr. Peter Small (the Investigator). The study will run until thirty (30) participants have completed the study

The Primary objective is to assess the agreement in cough counting between the Hyfe Cough Monitoring System and human listeners on an hour by hour basis when used by individuals with problematic cough under common living conditions using a Bland-Altman analysis.

The Hyfe Watch, along with the companion app, is part of the Hyfe Cough Monitoring System. It does not compromise the users provacy as it only retains the time of day associated with each cough. When the system detects a short explosive sound, it runs a brief "snippet" of that sound through a cough detection algorithm on the watch. If the algorithm deems the sound to be a cough, the device records the exact time that the cough occurred, and sends this time stamp to the companion app. The companion app does not access any personal information on the phone and is only used to "collect" the times at which a participant coughed from the Hyfe Watch and send them digitally to the researcher.

At the end of the 24 hours monitoring period envisiones, participants will be contacted by video call and asked to download this information from the companion app and send this to the Investigator. The use of the Hyfe Cough Monitoring System will not lead to additional medical interventions or changes to medical care.

In contrast, the sound recording watch will record all ambient sounds during a 24 hour period. This is necessary for the investigator to get an independent count of a participant´s coughing. As such, the sound recording watch will record conversations and those in the participant´s environment during this 24 hour period. It is important to let others in the environment know that sound is being recorded. The recordings will not be directly linked with the participant´s identity and will only be listened to by researchers who are trained in how to ensure the privacy of this data.

The data collected from the sound recording watch will NOT be transferred through the internet while participants are wearing it. Audio recordings will be saved on the actual device. Investigators will download the audio recordings onto a computer after the return the devices. Recordings will then be fully deleted.

Criteria for success:

The goal of this study is to demonstrate the performance of the Hyfe Cough Monitoring System as a device that continually and unobtrusively monitors cough. As has been agreed upon with the FDA, There is no pre-specified performance goal for the HCMS, this information will be reported in the labeling material. Therefore, the success of this study will be judged based on demonstrating adequate precision of our endpoints as quantified by their margin of error. Thus, the study will be considered satisfactory if the following criteria are satisfied:

Bland-Altman analysis:

* The bootstrap confidence interval for the bias has endpoints of magnitude at most 0.5.
* The endpoints of the bootstrap confidence intervals surrounding the 95% Limits of Agreement have magnitude at most 5.
* The regression line fitting the Bland-Altman plot has a slope that does not differ significantly from 0. This will confirm that the hourly differences do not suffer from proportional bias.

These 95% Bland-Altman Limits of Agreement (LOA) criteria correspond to the extreme acceptable differences between Hyfe's cough-second counts and those of human annotators; by requiring these limits to have magnitude at most 5, it is expected that most of the differences to have magnitude less than 5. Note that the accompanying criterion for success for the bias is that its confidence interval have endpoints of magnitude at most 0.5, so it is expected that the average difference to be close to 0.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Have problematic cough defined as an expressed concern about their cough
* Able to collect 24 hour auditory recording
* Reside in location without unusually high noise
* Willing to wear watches for 24 hours
* Fluent in English
* Access to a device for video calls
* Have an iPhone for download of the Hyfe Companion App
* Accept the Hyfe Companion App Terms of Use and Privacy Policy

Exclusion Criteria:

* Ongoing relationship with any company making a cough monitor
* Participation in a cough monitor device study in the past 6 months
* Have privacy concerns
* Inability to avoid unusually loud environments
* Significant antitussive therapy changes in preceding week

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects residing in the United States who have problematic coughs due to a variety of etiologies who are willing and able to participate in a decentralized study
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Hour by hour cough count agreement using Bland Altman | 24 hours
  Concordance with human annotators using Bland Altman analysis with 95%CI

SECONDARY OUTCOMES:
Hour by hour cough count agreement using linear analysis | 24 hours
  Concordance with human annotators using linear analysis
Event by event cough count analysis | 24 hours
  Agreement with human anotators in terms of sensitivity, false positive rate and positive predictive value

OTHER OUTCOMES:
Differential performance of Hyfe day/night | 24 hours
  Using Bland Altman Linear analysis Sensitivity, false positive rate and positive predictive value
Differential performance of Hyfe between individuals | 24 hours
  Using Bland Altman Linear analysis Sensitivity, false positive rate and positive predictive value
Differential performance of Hyfe between high, middle and low cough rates | 24 hours
  Using Bland Altman Linear analysis Sensitivity, false positive rate and positive predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Small, MD, Principal Investigator — Hyfe Inc
Locations (1):
- Hyfe. Inc, Ottawa, Montana, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified cough counts will be posted publicly in Hyfes GitHub repository
Supporting Information: Study Protocol
Time Frame: Within one year of study end
Access Criteria: Upon contacting the PI with reasonable request